CLINICAL TRIAL: NCT00842829
Title: A European Multicenter Open-Label Study of Breakthrough Cancer Pain: Assessment of Fentanyl Buccal Tablets Titration and Treatment in Opioid-Tolerant Patients
Brief Title: Study of Breakthrough Cancer Pain: Assessment of Fentanyl Buccal Tablets Titration and Treatment in Opioid-Tolerant Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment stopped at the end of the recruitment timeframe
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: C25608/4027/BP/EU; 2008-001841-24 (EudraCT Number)
Record Dates: First submitted 2009-01-29; First posted 2009-02-12 (Estimated); Results first posted 2012-09-20 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Cancer Pain; Breakthrough Pain
Keywords: Breakthrough Cancer Pain
MeSH Terms: conditions — Cancer Pain; Breakthrough Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FBT 100 mcg (Experimental): During the Titration Period, participants took fentanyl buccal tables (FBT) with a starting dose of 100 mcg until they reached an effective dose, with a maximum dose of 800 mcg and a maximum timeframe of 7 days. Participants who reached an effective dose entered the Open-label Treatment Period, whose length depended on how long was needed to treat up to 8 episodes of breakthrough pain (BTP) with FBT (maximum of 8 days). The length of the Continuation Period (when applicable) varied from country to country, up to until FBT was commercially available in that country.
  Interventions: Drug: Fentanyl Buccal Tablet (FBT)
- FBT 200 mcg (Active Comparator): During the Titration Period, participants took fentanyl buccal tables (FBT) with a starting dose of 200 mcg until they reached an effective dose, with a maximum dose of 800 mcg and a maximum timeframe of 7 days. Participants who reached an effective dose entered the Open-label Treatment Period, whose length depended on how long was needed to treat up to 8 episodes of breakthrough pain (BTP) with FBT (maximum of 8 days). The length of the Continuation Period (when applicable) varied from country to country, up to until FBT was commercially available in that country.
  Interventions: Drug: Fentanyl Buccal Tablet (FBT)

INTERVENTIONS:
Drug: Fentanyl Buccal Tablet (FBT) — FBTs were self-administered by participants via the oral mucosa. During the open-label dose titration period, participants used 1 to 4 tablets of the 100 mcg or 200 mcg strength to individually titrate upwards to an effective dose through the range of available strengths (i.e. 100, 200, 400, 600, or 800 mcg). For the open-label treatment and continuation periods, single dose tablets at the effective dose identified during the titration period were used. The maximum dose allowed per breakthrough pain (BTP) episode was 800 mcg. On any single day, participants were not to use FBT for more than 4 BTP episodes.
  Other Names: Fentora; CEP-25608; Fentanyl citrate; Effentora

SUMMARY:
Breakthrough cancer pain (BTcP) is a common problem in patients with cancer. Fentanyl Buccal Tablet (FBT) is used for the treatment of BTP in adults with cancer who are already receiving maintenance opioid therapy for chronic cancer pain. FBT treatment should be individually titrated to an effective dose that provides adequate analgesia and minimizes undesirable effects. To reach the safest effective dose for the individual patient as soon as possible, the dose titration process is critical. The aim of this study, conducted under pragmatic conditions in a large-scale population of cancer patients is to compare the proportion of patients reaching an effective FBT dose after titration starting with either a 100 mcg dose or a 200 mcg dose.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing to provide written informed consent to participate in this study.
* The patient can be either an out-patient or an in-patient.
* The patient has a histologically documented diagnosis of cancer.
* The patient has stable background pain due to cancer.
* The patient experiences up to 4 BTcP episodes per 24 hours.
* As maintenance opioid therapy, the patient is currently taking 1 of the following: at least 60 mg of oral morphine/day, at least 25 mcg of transdermal fentanyl/hour, at least 30 mg of oxycodone/day, at least 8 mg of hydromorphone/day, of an equianalgesic dose of another opioid for a week or longer before administration of the first dose of study drug.
* Women of childbearing potential, using a medically accepted, highly effective method of birth control and agree to continued use of this method for the duration of the study.
* The patient must be willing and able to successfully self-administer the study drug and to fill in study documents.

Exclusion Criteria:

* The patient is without maintenance opioid therapy.
* The patient has uncontrolled or rapidly escalating pain as determined by the investigator.
* The patient has known or suspected hypersensitivities, allergies, or other contraindications to the active drug or to any of the excipients of the study drug.
* The patient has respiratory depression or chronic obstructive pulmonary disease, or any other medical condition predisposing to respiratory depression.
* The patient has medical or psychiatric disease that, in the opinion of the investigator, would compromise collected data.
* The patient is expected to have surgery during the study.
* The patient is pregnant or lactating.
* The patient has participated in a study involving an investigational drug in the prior 30 days.
* The patient has received a monoamine oxidase inhibitor (MAOI) within 14 days before the first treatment with study drug.
* The patient has any other medical condition or is receiving concomitant medication/therapy (e.g., regional nerve block) that could, in the opinion of the investigator, compromise the patient's safety or compliance with the study protocol, or compromise collected data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon Europe
Locations (104):
- France (20):
  - Investigational Site, Bayonne
  - Investigational Site, Bordeaux
  - Investigational Site, Caen
  - Investigational Site, Clichy
  - Investigational Site, Grenoble
  - Investigational Site, Le Chesnay
  - Investigational Site, Le Kremlin-Bicêtre
  - Investigational Site, Le Mans
  - Investigational Site, Lorient
  - Investigational Site, Montpellier
  - Investigational Site, Nevers
  - Investigational Site, Orléans
  - Investigational Site, Paris
  - Investigational Site, Pierre-Bénite
  - Investigational Site, Poitiers
  - Investigational Site, Rouen
  - Investigational Site, Saint-Herblain
  - Investigational Site, Tarbes
  - Investigational Site, Toulouse
  - Investigational Site, Villejuif
- Germany (26):
  - Investigational Site, Bad Honnef
  - Investigational Site, Bad Lippspringe
  - Investigational Site, Berlin
  - Investigational Site, Bonn
  - Investigational Site, Böhlen
  - Investigational Site, Dresden
  - Investigational Site, Duisburg
  - Investigational Site, Erfurt
  - Investigational Site, Freiburg im Breisgau
  - Investigational Site, Geesthacht
  - Investigational Site, Greifenstein
  - Investigational Site, Hanover
  - Investigational Site, Herne
  - Investigational Site, Hildesheim
  - Investigational Site, Jena
  - Investigational Site, Kassel
  - Investigational Site, Leipzig
  - Investigational Site, Lohsa
  - Investigational Site, Lünen
  - Investigational Site, Mainz
  - Investigational Site, Munich
  - Investigational Site, Mülhausen
  - Investigational Site, Neustadt
  - Investigational Site, Rostock
  - Investigational Site, Weiden
  - Investigational Site, Würselen
- Investigational Site, Dublin, Ireland
- Italy (21):
  - Investigational Site, Aviano
  - Investigational Site, Bari
  - Investigational Site, Brescia
  - Investigational Site, Cagliari
  - Investigational Site, Candiolo
  - Investigational Site, Caserta
  - Investigational Site, Cosenza
  - Investigational Site, Florence
  - Investigational Site, Garbagnate Milanese
  - Investigational Site, Genova
  - Investigational Site, Lugo
  - Investigational Site, L’Aquila
  - Investigational Site, Milan
  - Investigational Site, Modena
  - Investigational Site, Napoli
  - Investigational Site, Palermo
  - Investigational Site, Piacenza
  - Investigational Site, Pisa
  - Investigational Site, Roma
  - Investigational Site, Torino
  - Investigational Site, Verona
- Poland (13):
  - Investigational Site, Bielsko-Biala
  - Investigational Site, Bydgoszcz
  - Investigational Site, Elblag
  - Investigational Site, Gdansk
  - Investigational Site, Gliwice
  - Investigational Site, Lodz
  - Investigational Site, Poznan
  - Investigational Site, Puszczykowo
  - Investigational Site, Szczecin
  - Investigational Site, Tychy
  - Investigational Site, Warsaw
  - Investigational Site, Wroclaw
  - Investigational Site, Włocławek
- Spain (16):
  - Investigational Site, A Coruña
  - Investigational Site, Barcelona
  - Investigational Site, Bilbao
  - Investigational Site, Cadiz
  - Investigational Site, Córdoba
  - Investigational Site, Granada
  - Investigational Site, Lleida
  - Investigational Site, Madrid
  - Investigational Site, Palma de Mallorca
  - Investigational Site, Pamplona
  - Investigational Site, Salamanca
  - Investigational Site, San Cristóbal de La Laguna
  - Investigational Site, Santander
  - Investigational Site, Santiago de Compostela
  - Investigational Site, Seville
  - Investigational Site, Valencia
- United Kingdom (7):
  - Investigational Site, Bath
  - Investigational Site, Dumfries
  - Investigational Site, London
  - Investigational Site, Nottingham
  - Investigational Site, Plymouth
  - Investigational Site, Surrey
  - Investigational Site, Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 442 patients already receiving opioid maintenance therapy for chronic cancer pain and experiencing up to 4 BTP episodes per 24 hours (on average) were screened at 135 centers in 7 European countries.
Groups:
- FBT 100 Mcg - Dose Titration Period: During the Titration Period, participants took fentanyl buccal tables (FBT) with a starting dose of 100 mcg until they reached an effective dose, with a maximum dose of 800 mcg and a maximum timeframe of 7 days.
- FBT 200 Mcg - Dose Titration Period: During the Titration Period, participants took fentanyl buccal tables (FBT) with a starting dose of 200 mcg until they reached an effective dose, with a maximum dose of 800 mcg and a maximum timeframe of 7 days.
- FBT - Treatment and Continuation Periods: Participants who reached an effective dose entered the Open-label Treatment Period, whose length depended on how long was needed to treat up to 8 episodes of breakthrough pain (BTP) with FBT (maximum of 8 days). The length of the Continuation Period (when applicable) varied from country to country, up to until FBT was commercially available in that country.
Period: Dose Titration Period
Arm/Group | FBT 100 Mcg - Dose Titration Period | FBT 200 Mcg - Dose Titration Period | FBT - Treatment and Continuation Periods
Started | 156 | 174 | 0
Titration Safety Analysis Set | 145 (Received at least one dose of study drug) | 167 (Received at least one dose of study drug) | 0
Completed | 130 | 151 | 0
Not Completed | 26 | 23 | 0
Not completed — Adverse Event | 11 | 10 | 0
Not completed — Lack of Efficacy | 4 | 1 | 0
Not completed — Unstable persistent cancer pain | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 6 | 0
Not completed — Other | 5 | 4 | 0
Not completed — Non-compliance to study procedures | 1 | 1 | 0
Not completed — Non-compliance to study drug | 2 | 1 | 0
Period: Treatment Period
Arm/Group | FBT 100 Mcg - Dose Titration Period | FBT 200 Mcg - Dose Titration Period | FBT - Treatment and Continuation Periods
Started | 0 | 0 | 281
Safety Analysis Set | 0 | 0 | 223 (Received at least one dose of study drug)
Completed | 0 | 0 | 218
Not Completed | 0 | 0 | 63
Not completed — Adverse Event | 0 | 0 | 15
Not completed — Lack of Efficacy | 0 | 0 | 6
Not completed — Unstable persistent cancer pain | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 11
Not completed — Consistently >4 BTP episodes daily | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Other | 0 | 0 | 18
Not completed — Non-compliance to study procedures | 0 | 0 | 4
Not completed — Unclear completion status | 0 | 0 | 1
Period: Continuation Period
Arm/Group | FBT 100 Mcg - Dose Titration Period | FBT 200 Mcg - Dose Titration Period | FBT - Treatment and Continuation Periods
Started | 0 | 0 | 88 (Eligible for Continuation Period)
Continuation Safety Analysis Set | 0 | 0 | 87 (Received at least one dose of study drug)
Completed | 0 | 0 | 27
Not Completed | 0 | 0 | 61
Not completed — Adverse Event | 0 | 0 | 32
Not completed — Lack of Efficacy | 0 | 0 | 6
Not completed — Unstable persistent cancer pain | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 10
Not completed — Other | 0 | 0 | 7
Not completed — Non-compliance to study procedures | 0 | 0 | 2
Not completed — Non-compliance to study drug | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FBT 100 Mcg - Dose Titration Period | FBT 200 Mcg - Dose Titration Period | Total
Number analyzed (Participants) | 156 | 174 | 330
Age Continuous [Mean (Standard Deviation); unit: years] | 59.5 (11.72) | 60.1 (10.97) | 59.8 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 78 | 149
  Male | 85 | 96 | 181
Region of Enrollment [Number; unit: participants]
  France | 16 | 25 | 41
  Spain | 26 | 26 | 52
  Poland | 38 | 41 | 79
  Ireland | 1 | 0 | 1
  Germany | 32 | 38 | 70
  United Kingdom | 8 | 7 | 15
  Italy | 35 | 37 | 72
Cancer Site [Number; unit: participants]
  Breast | 31 | 36 | 67
  Colon/rectum | 15 | 25 | 40
  Colon/rectum + Pancreas/stomach + other | 1 | 0 | 1
  Head/neck | 12 | 12 | 24
  Leukemia/lymphoma | 2 | 4 | 6
  Myeloma | 5 | 4 | 9
  Oesophageal | 4 | 2 | 6
  Pancreas/stomach | 13 | 11 | 24
  Prostate | 8 | 17 | 25
  Lung | 26 | 21 | 47
  Other (not specified) | 39 | 42 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reaching an Effective Fentanyl Buccal Tablet (FBT) Dose As Assessed by the Participant During the Titration Period
Description: The effective dose was the dose that, for 2 consecutive break-through pain (BTP) episodes, provided adequate analgesia within the first 30 minutes after administration of study drug and that minimized undesirable effects. The assessment was performed by the participant and was reported in the titration-period diary. The next BTP episode was used to confirm the effective dose, and if confirmed, the effective dose was used for all following BTP episodes.
Time Frame: Day 1 up to Day 7
Population: Titration safety analysis set consisting of participants who took at least one dose of study medication.
Measure: Number; unit: percentage of treated participants
Arm/Group | FBT 100 Mcg - Dose Titration Period | FBT 200 Mcg - Dose Titration Period
Number analyzed (Participants) | 145 | 167
percentage of treated participants | 75.2 | 81.2
Statistical Analysis 1: Comparison: FBT 100 Mcg - Dose Titration Period vs FBT 200 Mcg - Dose Titration Period; Treatment comparison difference (100 mcg - 200 mcg); Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the upper limit of the 90% CI was <8%; Mean Difference (Net) = -6.3, 95% CI 1-sided [upper limit 1.4] — The upper bound of the 2-sided 90% confidence interval is equivalent to the upper bound of the 1-sided 95% confidence interval

2. Secondary Outcome: Kaplan-Meier Estimates for Time to Meaningful Pain Relief As Assessed by Participants During the Treatment Period For Overall Breakthrough Pain (BTP) Episodes
Description: Overall episode data analyzed all values of time to meaningful pain relief taken over all BTP episodes during the treatment period. If meaningful pain relief was not achieved within 60 minutes of FBT intake, or if rescue medication was taken, the event was censored. Meaningful pain relief was left to the judgment of participants, who used a stopwatch and recorded the time from treatment until pain relief in a patient diary.
Time Frame: approximately Day 8-15
Population: Safety analysis set consisting of participants who received at least one dose of study drug during the Treatment Period, and who recorded the time to pain relief in the patient diary.
Measure: Median (Inter-Quartile Range); unit: minutes
Units Other Than Participants: breakthrough pain episodes
Groups:
- FBT - Treatment Period: Participants who reached an effective dose entered the Open-label Treatment Period, whose length depended on how long was needed to treat up to 8 episodes of breakthrough pain (BTP) with FBT (maximum of 8 days).
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 214
Number analyzed (breakthrough pain episodes) | 1810
minutes | 19.00 [12.00 to 30.00]

3. Secondary Outcome: Number of Participants Reaching An Effective Dose As Assessed by the Participant During the Titration Period
Description: Number of participants for which an effective dose of FBT was reached as judged by each participant. The effective dose was the dose that, for 2 consecutive break-through pain (BTP) episodes, provided adequate analgesia within the first 30 minutes after administration of study drug and that minimized undesirable effects. The assessment was performed by the participant and was reported in the titration-period diary. The next BTP episode was used to confirm the effective dose, and if confirmed, the effective dose was used for all following BTP episodes.
Time Frame: Day 1 up to Day 7
Population: Titration safety analysis set consisting of participants who took at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | FBT 100 Mcg - Dose Titration Period | FBT 200 Mcg - Dose Titration Period
Number analyzed (Participants) | 145 | 167
participants
  100 mcg | 34 | 7
  200 mcg | 38 | 61
  300 mcg (evaluated by mistake) | 1 | 1
  400 mcg | 23 | 42
  600 mcg | 8 | 15
  800 mcg | 5 | 10
  Missing | 36 | 31

4. Secondary Outcome: Breakthrough Pain (BTP) Episodes Requiring the Use of Rescue Medication During the Titration Period and the Treatment Period
Description: The number of breakthrough pain (BTP) episodes in which the participant did not obtain effective pain relief from study medication and took a rescue medication.
Time Frame: Days 1 to up to Day 7 (Titration Period); approximately Day 8 up to Day 15 (Treatment Period)
Population: Safety analysis set consisting of participants who took at least one dose of study drug during the relevant study period.
Measure: Number; unit: BTP episodes
Units Other Than Participants: breakthrough pain episodes
Groups:
- During Titration Period: The titration period consisted of up to 7 days of treatment in which participants used increasing dosage of study drug in order to identify the effective dose for their breakthrough pain episodes.
- During Treatment Period: The treatment period included participants who identified an effective dose during the earlier study period and used that dose for BTP episodes during the Treatment Period.
Arm/Group | During Titration Period | During Treatment Period
Number analyzed (Participants) | 223 | 223
Number analyzed (breakthrough pain episodes) | 2610 | 1810
BTP episodes | 102 | 153

5. Secondary Outcome: Participant Assessment of Medication Performance During the Treatment Period
Description: Participants assessed the performance of FBT at 30 minutes and 60 minutes after dosing each episode during the treatment period. For each episode, the participant answered the question 'How well did your study medication perform in controlling the breakthrough pain episode?' on a 5-point Likert-type scale (poor=0, fair=1, good=2, very good=3, and excellent=4).
Time Frame: approximately Day 8-15
Population: Safety analysis set of participants with a response at the time point (30 or 60 minutes) post dose.
Measure: Number; unit: BTP episodes
Units Other Than Participants: breakthrough pain episodes
Groups:
- 30 Minutes: Participant assessments of medication performance 30 minutes after dosing during the Treatment Period.
- 60 Minutes: Participant assessments of medication performance 60 minutes after dosing during the Treatment Period.
Arm/Group | 30 Minutes | 60 Minutes
Number analyzed (Participants) | 222 | 214
Number analyzed (breakthrough pain episodes) | 1776 | 1668
BTP episodes
  Excellent | 103 | 144
  Very good | 433 | 584
  Good | 712 | 646
  Fair | 428 | 245
  Poor | 100 | 49
  Missing | 35 | 143

6. Secondary Outcome: Change From Baseline to End of Treatment Period (Approximately Day 15) in the Brief Pain Inventory 7-item (BPI-7S) Questionnaire Subscale: General Activity
Description: Participants completed the BPI-7S questionnaire to indicate their quality of life and functional status between study time points. For each subscale, the participant rated their responses from 0=Does not interfere through to 10=Completely interferes. A negative change from baseline represents an improvement.
  This subscale assesses general activity.
Time Frame: Day 0 (baseline), approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with both baseline and Treatment Period responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 206
units on a scale | -1.0 (2.52)

7. Secondary Outcome: Change From Baseline to End of Treatment Period (Approximately Day 15) in the Brief Pain Inventory 7-item (BPI-7S) Questionnaire Subscale: Mood
Description: Participants completed the BPI-7S questionnaire to indicate their quality of life and functional status between study time points. For each subscale, the participant rated their responses from 0=Does not interfere through to 10=Completely interferes. A negative change from baseline represents an improvement.
  This subscale assesses mood.
Time Frame: Day 0 (baseline), approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with both baseline and Treatment Period responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 205
units on a scale | -1.4 (2.55)

8. Secondary Outcome: Change From Baseline to End of Treatment Period (Approximately Day 15) in the Brief Pain Inventory 7-item (BPI-7S) Questionnaire Subscale: Walking Ability
Description: Participants completed the BPI-7S questionnaire to indicate their quality of life and functional status between study time points. For each subscale, the participant rated their responses from 0=Does not interfere through to 10=Completely interferes. A negative change from baseline represents an improvement.
  This subscale assesses walking ability.
Time Frame: Day 0 (baseline), approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with both baseline and Treatment Period responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 201
units on a scale | -0.9 (2.29)

9. Secondary Outcome: Change From Baseline to End of Treatment Period (Approximately Day 15) in the Brief Pain Inventory 7-item (BPI-7S) Questionnaire Subscale: Normal Work
Description: Participants completed the BPI-7S questionnaire to indicate their quality of life and functional status between study time points. For each subscale, the participant rated their responses from 0=Does not interfere through to 10=Completely interferes. A negative change from baseline represents an improvement.
  This subscale assesses normal work.
Time Frame: Day 0 (baseline), approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with both baseline and Treatment Period responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 200
units on a scale | -1.3 (2.61)

10. Secondary Outcome: Change From Baseline to End of Treatment Period (Approximately Day 15) in the Brief Pain Inventory 7-item (BPI-7S) Questionnaire Subscale: Relations With Other People
Description: Participants completed the BPI-7S questionnaire to indicate their quality of life and functional status between study time points. For each subscale, the participant rated their responses from 0=Does not interfere through to 10=Completely interferes. A negative change from baseline represents an improvement.
  This subscale assesses relations with other people.
Time Frame: Day 0 (baseline), approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with both baseline and Treatment Period responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 205
units on a scale | -1.2 (2.50)

11. Secondary Outcome: Change From Baseline to End of Treatment Period (Approximately Day 15) in the Brief Pain Inventory 7-item (BPI-7S) Questionnaire Subscale: Sleep
Description: Participants completed the BPI-7S questionnaire to indicate their quality of life and functional status between study time points. For each subscale, the participant rated their responses from 0=Does not interfere through to 10=Completely interferes. A negative change from baseline represents an improvement.
  This subscale assesses sleep.
Time Frame: Day 0 (baseline), approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with both baseline and Treatment Period responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 204
units on a scale | -1.4 (2.66)

12. Secondary Outcome: Change From Baseline to End of Treatment Period (Approximately Day 15) in the Brief Pain Inventory 7-item (BPI-7S) Questionnaire Subscale: Enjoyment of Life
Description: Participants completed the BPI-7S questionnaire to indicate their quality of life and functional status between study time points. For each subscale, the participant rated their responses from 0=Does not interfere through to 10=Completely interferes. A negative change from baseline represents an improvement.
  This subscale assesses enjoyment of life.
Time Frame: Day 0 (baseline), approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with both baseline and Treatment Period responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 204
units on a scale | -1.5 (2.77)

13. Secondary Outcome: Change From Baseline to End of Treatment Period (Approximately Day 15) in the Brief Pain Inventory 7-item (BPI-7S) Questionnaire: Global Score
Description: Participants completed the BPI-7S questionnaire to indicate their quality of life and functional status between study time points. For each subscale, the participant rated their responses from 0=Does not interfere through to 10=Completely interferes. The Global Score is the sum of the subscales (total scale is 0-70). A negative change from baseline represents an improvement.
Time Frame: Day 0 (baseline), approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with both baseline and Treatment Period responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 198
units on a scale | -8.6 (13.47)

14. Secondary Outcome: Participant's Global Assessment of Satisfaction (Satisfied With BTP Treatment?) at the End of the Treatment Period
Description: Responses to the Patient Satisfaction questionnaire question, "Satisfied with the BTP Treatment?", were captured on a five-point scale from 0=not at all to 4=very much.
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 203
participants
  Very much | 64
  Quite a bit | 92
  Somewhat | 37
  A little bit | 8
  Not at all | 2

15. Secondary Outcome: Participant's Global Assessment of Satisfaction (Does This BTP Medication Relieve Your Pain Quickly so You Can Get Back to Sleep?) at the End of the Treatment Period
Description: Responses to the Patient Satisfaction questionnaire question, "Does this BTP medication relieve your pain quickly so you can get back to sleep?", were captured on a five-point scale from 0=not at all to 4=very much.
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 202
participants
  Very much | 55
  Quite a bit | 104
  Somewhat | 27
  A little bit | 13
  Not at all | 3

16. Secondary Outcome: Participant's Global Assessment of Satisfaction (Does This Medication Work Fast?) at the End of the Treatment Period
Description: Responses to the Patient Satisfaction questionnaire question, "Does this medication work fast?", were captured on a five-point scale from 0=not at all to 4=very much.
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 203
participants
  Very much | 63
  Quite a bit | 88
  Somewhat | 36
  A little bit | 12
  Not at all | 4

17. Secondary Outcome: Participant's Global Assessment of Satisfaction (Does This Medication Provide Adequate Relief?) at the End of the Treatment Period
Description: Responses to the Patient Satisfaction questionnaire question, "Does this medication provide adequate relief?", were captured on a five-point scale from 0=not at all to 4=very much.
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 203
participants
  Very much | 57
  Quite a bit | 104
  Somewhat | 35
  A little bit | 5
  Not at all | 2

18. Secondary Outcome: Participant's Global Assessment of Satisfaction (Is This Medication Easy to Take?) at the End of the Treatment Period
Description: Responses to the Patient Satisfaction questionnaire question, "Is this medication easy to take?", were captured on a five-point scale from 0=not at all to 4=very much.
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 203
participants
  Very much | 81
  Quite a bit | 74
  Somewhat | 31
  A little bit | 9
  Not at all | 8

19. Secondary Outcome: Participant's Global Assessment of Satisfaction (Do You Find This Medication Comfortable to Take in Public?) at the End of the Treatment Period
Description: Responses to the Patient Satisfaction questionnaire question, "Do you find this medication comfortable to take in public?", were captured on a five-point scale from 0=not at all to 4=very much.
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 203
participants
  Very much | 81
  Quite a bit | 78
  Somewhat | 26
  A little bit | 10
  Not at all | 8

20. Secondary Outcome: Participant's Global Assessment of Satisfaction (Do You Feel Safe Taking This Medication?) at the End of the Treatment Period
Description: Responses to the Patient Satisfaction questionnaire question, "Do you feel safe taking this medication?", were captured on a five-point scale from 0=not at all to 4=very much.
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 203
participants
  Very much | 96
  Quite a bit | 88
  Somewhat | 17
  A little bit | 2
  Not at all | 0

21. Secondary Outcome: Participant's Global Assessment of Satisfaction (Do You Understand the Instructions?) at the End of the Treatment Period
Description: Responses to the Patient Satisfaction questionnaire question, "Do you understand the instructions?", were captured on a five-point scale from 0=not at all to 4=very much.
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 203
participants
  Very much | 107
  Quite a bit | 81
  Somewhat | 13
  A little bit | 2
  Not at all | 0

22. Secondary Outcome: Participant's Global Assessment of Ease of Use at the End of the Treatment Period
Description: Ease of use was assessed using the question 'Did you find this treatment easy/convenient to use for treatment of your breakthrough pain episodes?'. The answer was based on a 4-point numerical scale (0=Poor, 1=Fair, 2=Easy, 3=Very Easy). This assessment was performed at the end of the Treatment Period (or early termination).
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 209
participants
  Very easy | 67
  Easy | 107
  Fair | 28
  Poor | 7

23. Secondary Outcome: Participant's Global Impression of Change at the End of the Treatment Period
Description: Global impression of change was assessed using the question 'Since the start of the study, my overall status is?'. The answer was based on a 7-point scale (1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very much worse). This assessment was performed at the end of the Treatment Period (or early termination).
Time Frame: approximately Day 15 (end of Treatment Period)
Population: Safety analysis set of participants with a response
Measure: Number; unit: participants
Arm/Group | FBT - Treatment Period
Number analyzed (Participants) | 208
participants
  Very much improved | 15
  Much improved | 75
  Minimally improved | 65
  No change | 32
  Minimally worse | 14
  Much worse | 7
  Very much worse | 0

24. Secondary Outcome: Participants With Adverse Events (AE) Summarized by Treatment Period
Description: Participants with treatment-emergent adverse events are summarized by each treatment period. Relation to study drug was assessed by the investigator. The 'Any AE' category below includes serious adverse events.
Time Frame: Day 1-7 (Titration Period). Day 8-15 (Treatment Period), Days 16-688 (Continuation Period)
Population: Safety analysis set
Measure: Number; unit: participants
Groups:
- FBT - Continuation Period: The length of the Continuation Period (when applicable) varied from country to country, up to until FBT was commercially available in that country.
Arm/Group | FBT 100 Mcg - Dose Titration Period | FBT 200 Mcg - Dose Titration Period | FBT - Treatment Period | FBT - Continuation Period
Number analyzed (Participants) | 145 | 167 | 223 | 87
participants
  Any AE | 44 | 74 | 43 | 72
  Any Serious AE | 8 | 12 | 4 | 37
  AE leading to discontinuation of study drug | 11 | 19 | 0 | 25
  AE with a fatal outcome | 6 | 4 | 3 | 29
  AE considered related to study drug | 19 | 35 | 15 | 14

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs from Day 1 up to day 688
Groups:
- FBT - All Doses and Study Periods: Participants took fentanyl buccal tables (FBT) with doses between 100-800 mcg
Arm/Group | FBT - All Doses and Study Periods
Serious Adverse Events (participants affected / at risk) | 67/312
Other Adverse Events (participants affected / at risk) | 52/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FBT - All Doses and Study Periods (N=312)
Anaemia (Blood and lymphatic system disorders) | 3
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 1
Cardiovascular insufficiency (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Tachycardia paroxysmal (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Oedema mouth (Gastrointestinal disorders) | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Tongue oedema (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Cyst (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Fatigue (General disorders) | 1
Feeling abnormal (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Infected cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Drug toxicity (Injury, poisoning and procedural complications) | 1
Cachexia (Metabolism and nutrition disorders) | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraparesis (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Superior vena caval occlusion (Vascular disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FBT - All Doses and Study Periods (N=312)
Nausea (Gastrointestinal disorders) | 30
Vomiting (Gastrointestinal disorders) | 23
Somnolence (Nervous system disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.